CLINICAL TRIAL: NCT03325101
Title: Phase Ib/II Study of Autologous Dendritic Cell Therapy Delivered Intratumorally After Cryoablation in Combination With Pembrolizumab for Patients With Metastatic or Unresectable Melanoma
Brief Title: Dendritic Cell Therapy With Pembrolizumab for Metastatic or Unresectable Melanoma
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: poor accrual
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: MC1771; NCI-2017-01967 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); MC1771 (Other: Mayo Clinic); 17-001666 (Other: Mayo Clinic Institutional Review Board)
Record Dates: First submitted 2017-10-25; First posted 2017-10-30 (Actual); Results first posted 2025-06-12 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2024-08

CONDITIONS: Stage III Cutaneous Melanoma AJCC v7; Stage IIIA Cutaneous Melanoma AJCC v7; Stage IIIB Cutaneous Melanoma AJCC v7; Stage IIIC Cutaneous Melanoma AJCC v7; Stage IV Cutaneous Melanoma AJCC v6 and v7
MeSH Terms: conditions — Melanoma | interventions — Cryosurgery; pembrolizumab; Blood Component Removal

STUDY DESIGN:
Intervention Model Description: Group 1: Phase I Schedule 1 Group 2: Phase I Schedule -1 (if Phase 1 Schedule 1 not well tolerated) Group 3: Phase II Schedule base on the findings of the Phase I portion of the trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Phase I Schedule 1 (Experimental): Phase I Schedule 1: Cycle length is 21 days with the exception of cycle 1 which may be extended an additional 7 days to allow for dendritic cell production.
  Cycle 1 Day 1: Patients undergo apheresis over 4 hours and pembrolizumab IV over 30 minutes.
  Cycle 2 & Cycle 3 Day 1: Pembrolizumab 200 mg is administered by IV over 30 minutes.
  Cycle 2 & Cycle 3 either Day 1 or Day 2 (within 36 hours of receiving pembrolizumab): patients undergo cryosurgery (injection of 30-60 x 10^6 mDCs and an injection of 0.5 ml Prenar13 such that two distinct metastatic lesions are cryoablated, one during cycle 2 and the other during cycle 3.
  Cycle 4 Day 1 and all subsequent cycles for a maximum of 2 years: Pembrolizumab 200 mg is administered by IV over 30 minutes
  Interventions: Procedure: Cryosurgery; Biological: Pembrolizumab; Procedure: Pheresis; Biological: Therapeutic Autologous Dendritic Cells
- Phase I Schedule -1 (Experimental): Phase I Schedule -1: Cycle length is 21 days with the exception of cycle 1 which may be extended an additional 7 days to allow for dendritic cell production.
  Cycle 1 Day 1: Patients undergo apheresis over 4 hours and pembrolizumab IV over 30 minutes.
  Cycle 2 & Cycle 3 either Day 1 or Day 2 (within 36 hours of receiving pembrolizumab): patients undergo cryosurgery (injection of 30-60 x 10^6 mDCs and an injection of 0.5 ml Prenar13 such that two distinct metastatic lesions are cryoablated, one during cycle 2 and the other during cycle 3.
  Cycle 4 Day 1 and all subsequent cycles for a maximum of 2 years: Pembrolizumab 200 mg is administered by IV over 30 minutes
  Interventions: Procedure: Cryosurgery; Biological: Pembrolizumab; Procedure: Pheresis; Biological: Therapeutic Autologous Dendritic Cells
- Phase II Schedule (Experimental): Regimen depends upon the results of the Phase I portion of the study.
  Interventions: Procedure: Cryosurgery; Biological: Pembrolizumab; Procedure: Pheresis; Biological: Therapeutic Autologous Dendritic Cells

INTERVENTIONS:
Procedure: Cryosurgery — Undergo cryosurgery
  Other Names: cryoablation; cryosurgical ablation
Biological: Pembrolizumab — IV
  Other Names: Keytruda; Lambrolizumab; MK-3475; SCH 900475
Procedure: Pheresis — apheresis
  Other Names: Apheresis; Blood Component Removal; Collection, Apheresis/Leukapheresis; Hemapheresis
Biological: Therapeutic Autologous Dendritic Cells — Intra-tumoral injection

SUMMARY:
This phase Ib/II trial studies how well dendritic cell therapy after cryosurgery in combination with pembrolizumab works in treating patients with stage III-IV melanoma that cannot be removed by surgery. Vaccines made from a person's white blood cells mixed with tumor proteins may help the body build an effective immune response to kill tumor cells. Cryosurgery, also known as cryoablation or cryotherapy, kills tumor cells by freezing them. Monoclonal antibodies, such as pembrolizumab, may block tumor growth in different ways by targeting certain cells. Giving dendritic cell therapy after cryosurgery in combination with pembrolizumab may work better in treating patients with melanoma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES OF PHASE I portion of the trial: To establish the safety and tolerability of the proposed treatment schedule in order to move it forward into the Phase II portion of the trial.

PRIMARY OBJECTIVES OF PHASE II portion of the trial:

I. To determine the objective response rate (ORR) of pembrolizumab combined with cryoablation and intratumoral mature dendritic cells (mDCs) in patients with metastatic melanoma that has failed to respond or has stopped responding to initial therapy with a PD-1 axis-blocking monoclonal antibody.

SECONDARY OBJECTIVES:

I. To assess the safety profile of pembrolizumab combined with cryoablation and intratumoral mDCs in patients with metastatic melanoma that have failed to respond or have stopped responding to initial therapy with a PD-1 axis-blocking monoclonal antibody.

II. To determine median progression-free survival (PFS) obtained with this approach in this patient population.

III. To determine median overall survival (OS) obtained with this approach in this patient population.

TERTIARY OBJECTIVES:

I. To quantitate tumor infiltrating lymphocytes (TILs) in tumor biopsies prior to and following cryoablation and intratumoral mDCs.

II. To measure PD-L1 levels in tumor biopsies and blood biopsies prior to and following cryoablation and to assess whether a change in PD-L1 levels differ among those patients who met the criteria for clinical benefit (progression-free and on study for at least 6 months) and those who do not.

III. To measure peripheral blood mononuclear cells (PBMC) proliferation and function after coculture with frozen tumor before and after intratumoral mDC injection.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed diagnosis of unresectable stage III or metastatic melanoma (stage IV) not amenable to curative local therapy
* Documented progression of disease after initiation of therapy with OR lack of response to therapy with a PD-1- or PD-L1-targeting monoclonal antibody (pembrolizumab, nivolumab, etc) after at least 18 weeks; NOTE: This treatment could have been at any time prior to registration
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0 or 1
* Minimum of 3 radiographically apparent lesions such that there is:

  * Minimum of one lesion in areas that have not been previously irradiated that is considered measurable by Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 criteria AND
  * Minimum of two lesions in areas that have not been previously irradiated that are determined by interventional radiology to be of a size and in a location that a single probe could ablate at least 75% of the lesion; Note: Hepatic lesions measuring =< 3 cm may be treated, as determined by interventional radiology; Note: Brain metastases are not acceptable as lesions defining measurable disease, nor are they candidate lesions for cryoablation
* Adequate venous access for apheresis as assessed by apheresis team; NOTE: If a central venous catheter is required for apheresis, the patient is not eligible
* Absolute neutrophil count (ANC) >= 1000/mm^3 obtained =< 14 days prior to registration
* Absolute lymphocyte count >= 500/mm^3 obtained =< 14 days prior to registration
* Platelet count >= 100,000/mm^3 obtained =< 14 days prior to registration
* Hemoglobin >= 10 g/dL obtained =< 14 days prior to registration
* Total bilirubin =< 1.5 x upper limit of normal (ULN), unless due to Gilbert?s disease obtained =< 14 days prior to registration
* Aspartate transaminase (AST)/serum glutamic-oxaloacetic transaminase (SGOT) and alanine transaminase (ALT)/serum glutamate pyruvate transaminase (SGPT) =< 2.5 x ULN obtained =< 14 days prior to registration
* Creatinine =< 1.5 x ULN or calculated creatinine clearance >= 60 mL/min for subject with creatinine ? 1.5 x institutional ULN obtained =< 14 days prior to registration
* Negative serum pregnancy test for persons of childbearing potential =< 7 days prior to registration
* Provide written informed consent
* Willing to return to the enrolling institution for follow-up (during active treatment and active monitoring phase of the study)
* Willing to provide tissue and blood samples for research purposes
* Willing to use adequate contraception while on the study and until 120 days after the last dose of study drug

Exclusion Criteria:

* Any of the following:

  * Pregnant persons
  * Nursing persons
* History of human immunodeficiency virus (HIV), hepatitis B, or hepatitis C
* Active tuberculosis or active, non-infectious pneumonitis
* Evidence of interstitial lung disease
* Active infection requiring the use of systemic antibiotics
* Symptomatic congestive heart failure (New York Heart Association classification III or IV cardiovascular disease, myocardial infarction =< 6 months prior to registration, unstable angina pectoris or cardiac arrhythmia =< 3 months prior to registration, or cardiac arrhythmia
* Currently receiving or have received any other investigational agent considered as a treatment for the primary neoplasm =< 21 days prior to registration
* History of other primary malignancy requiring systemic treatment =< 3 years prior to registration; patients must not be receiving chemotherapy or immunotherapy for another cancer; patients must not have another active malignancy requiring active treatment; EXCEPTIONS: Non-melanotic skin cancer or carcinoma-in-situ of the cervix
* Failure to recover from prior side effects of immune checkpoint inhibitor therapy to =< grade 1; NOTE: Patients will not be excluded for adrenal insufficiency or hypothyroidism secondary to immunotherapy provided they are receiving hormonal replacement
* Major surgery =< 4 weeks prior to registration
* Prior chemotherapy, targeted therapy, or radiation therapy =< 2 weeks prior to registration or who has not recovered (i.e. to =< grade 1 or baseline) from an adverse event due to the previously administered therapy
* History of hypersensitivity and anaphylactoid reactions to pneumococcal vaccine or any component of the formulation, including diphtheria toxoid
* Active autoimmune disease such as Crohn?s disease, rheumatoid arthritis, Sjogrens? disease, systemic lupus erythematosus, or similar conditions requiring systemic treatment within the past 3 months or a documented history of clinically severe autoimmune disease/syndrome difficult to control in the past; EXCEPTIONS (the following are allowed):

  * Vitiligo or resolved childhood asthma/atopy
  * Intermittent use of bronchodilators or local steroid injections
  * Hypothyroidism stable on hormone replacement
  * Diabetes stable with current management
  * History of positive Coombs test but no evidence of hemolysis
  * Psoriasis not requiring systemic treatment
  * Conditions not expected to recur in the absence of an external trigger
  * Secondary adrenal insufficiency from previous hypophysitis, currently on physiologic replacement steroid dosing only
* Coagulopathy, including the use of therapeutic anticoagulants that cannot be discontinued for the cryoablation procedure; NOTE: Heparin for line patency without detectable lab abnormalities for coagulation will be allowed
* Corticosteroid use =< 14 days prior to registration; NOTE: Patients must be off systemic corticosteroids for at least 2 weeks prior to registration; this includes oral or IV route of administration; patients on chronic corticosteroids for adrenal insufficiency or other reasons may enroll if they receive less than 10 mg/day of prednisone (or equivalent); patients receiving inhaled or intranasal or intra-articular steroids are not excluded
* Active central nervous system (CNS) metastasis; NOTE: Patients with prior brain metastases that are asymptomatic without corticosteroid use and stable or improved >= 90 days after treatment with surgery or radiation are not excluded
* Receipt of a live vaccine =< 30 days prior to registration

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2017-11-15 (Actual); Primary Completion 2020-06-14 (Actual); Study Completion 2020-06-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Matthew S. Block, M.D., Ph.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared with investigators following the policies and procedures of the Mayo Clinic Cancer Center.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Available for 10 years post study closure.

REFERENCES:
- See also: Mayo Clinic web site — https://www.mayoclinic.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This Phase I/II clinical trial was designed to identify a treatment schedule for pembrolizumab in combination with cryoablation and intra-tumoral injection of mature dendritic cells (mDCs) with an acceptable safety profile (Phase 1) and then to assess anti-tumor activity (Phase II). The trial opened to enrollment November 15, 2017. The trial closed due to poor accrual on July 21, 2021, having enrolled 7 pts onto Phase I Schedule 1 cohort. The final patient occurred June 14, 2020.
Groups:
- Treatment (Apheresis, Pembrolizumab, Cryosurgery, Mature Dendritic Cells [mDCs]): Phase I Schedule 1 Treatment cohort where cycle length is 21 days: On D1C1, patients undergo apheresis and receive 200mg pembrolizumab IV over 30 minutes. On C2D1, patients will receive 200 mg pembrolizumab administered IV over 30 minutes. Within 36 hours of receiving pembrolizumab, a single metastatic lesion will be biopsied and cryoablated (using conventional freeze-thaw-freeze cycle). After the lesion has thawed, a 22 G needle will be placed under ultrasound or CT-guidance into the ablated portion of the lesion. The mature Dendritic Cells (total mDCS: 30-60 x10^6) will be administered through this needle over different areas of the cryoablated region and then flushed with 1 ml of sterile saline. Prevnar13® will be injected into the ablated portion of the lesion after administration of mDCs. On C3D1 the same treatment will be administered to a different metastatic lesion. C4D1 and D1 of all subsequent cycle patients will receive 200 mg pembrolizumab IV over 30 minutes. Treatment continues until disease progression or a maximum of 24 months post registration
Period: Overall Study
Arm/Group | Treatment (Apheresis, Pembrolizumab, Cryosurgery, Mature Dendritic Cells [mDCs])
Started | 7
Completed | 7
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Study closed to enrollment due to poor accrual.
Groups:
- Phase I Schedule 1: Phase I Schedule 1 Treatment cohort where cycle length is 21 days: On D1C1, patients undergo apheresis and receive 200mg pembrolizumab IV over 30 minutes. On C2D1, patients will receive 200 mg pembrolizumab administered IV over 30 minutes. Within 36 hours of receiving pembrolizumab, a single metastatic lesion will be biopsied and cryoablated (using conventional freeze-thaw-freeze cycle). After the lesion has thawed, a 22 G needle will be placed under ultrasound or CT-guidance into the ablated portion of the lesion. The mature Dendritic Cells (total mDCS: 30-60 x10^6) will be administered through this needle over different areas of the cryoablated region and then flushed with 1ml of sterile saline. Prevnar13® will be injected into the ablated portion of the lesion after administration of mDCs. On C3D1 the same treatment will be administered to a different metastatic lesion. C4D1 and D1 of all subsequent cycle patients will receive 200mg pembrolizumab IV over 30 minutes. Treatment continues until disease progression or a maximum of 24 months post registration.
- Phase I Schedule -1: hase I Schedule 1 Treatment cohort where cycle length is 21 days: On D1C1, patients undergo apheresis and receive 200mg pembrolizumab IV over 30 minutes. On C2D1, a single metastatic lesion will be biopsied and cryoablated (using conventional freeze-thaw-freeze cycle). After the lesion has thawed, a 22 G needle will be placed under ultrasound or CT-guidance into the ablated portion of the lesion. The mature Dendritic Cells (total mDCS: 30-60 x10^6) will be administered through this needle over different areas of the cryoablated region and then flushed with 1ml of sterile saline. Prevnar13® will be injected into the ablated portion of the lesion after administration of mDCs. On C3D1 the same treatment will be administered to a different metastatic lesion. C4D1 and D1 of all subsequent cycle patients will receive 200mg pembrolizumab IV over 30 minutes. Treatment continues until disease progression or a maximum of 24 months post registration.
- Phase II Schedule: Phase II Schedule based on the findings of the Phase I portion of the study
- Total: Total of all reporting groups
Arm/Group | Phase I Schedule 1 | Phase I Schedule -1 | Phase II Schedule | Total
Number analyzed (Participants) | 7 | 0 | 0 | 7
Age, Customized [Median (Full Range); unit: years]
  Age at study entry | 65.4 [58.4 to 76.2] |  |  | 65.4 [58.4 to 76.2]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 |  |  | 2
  Male | 5 |  |  | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 |  |  | 0
  Not Hispanic or Latino | 7 |  |  | 7
  Unknown or Not Reported | 0 |  |  | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 |  |  | 0
  Asian | 0 |  |  | 0
  Native Hawaiian or Other Pacific Islander | 0 |  |  | 0
  Black or African American | 0 |  |  | 0
  White | 7 |  |  | 7
  More than one race | 0 |  |  | 0
  Unknown or Not Reported | 0 |  |  | 0
Region of Enrollment [Number; unit: participants]
  United States | 7 |  |  | 7
ECOG Performance Status at Study entry [Count of Participants; unit: Participants] — Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) is a measurement of how well a patient can manage daily activities and self-care. The scale ranges from 0 (fully active) to 5 (dead), with higher numbers indicating increasing disability and limitations in activity.
  Participants
    ECOG PS = 0 | 5 |  |  | 5
    ECOG PS = 1 | 2 |  |  | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Developed a DLT During the First 3 Cycles of Treatment.
Description: The primary outcome of the Phase I portion of this trial was to establish the tolerability of the proposed treatment schedule in order to move it forward into the Phase II portion of the trial. A maximum of 6 patients was to be enrolled onto the Schedule 1. If at most one of these 6 patients developed a DLT during the first 3 treatment cycles, then Schedule #1 would be carried forward to the Phase II portion of the trial. If not, then an additional 6 patients would be treated with a modified Schedule 1 where Pembrolizumab was eliminated from cycles 2 & 3. Dose-limiting toxicity (DLT) were defined as the following possibly, probably, or definitely related AEs to protocol therapy during first 3 treatment cycles: Grade 3+ infusion reactions, acute kidney injury, chronic kidney disease, pneumonitis; or Grade 2 infusion reactions, acute kidney injury, chronic kidney disease or pneumonitis that does not resolve to Grade 0-1 within 21 days.
Time Frame: Up to 3 months (3 cycles of 21 days and an additional 7 days for Cycle 1)
Population: All patient who began protocol treatment.
Measure: Count of Participants; unit: Participants
Groups:
- Phase I Schedule 1: Cycle length is 21 days with the exception of cycle 1 which may be extended an additional 7 days to allow for dendritic cell production
  Patients undergo apheresis over 4 hours and pembrolizumab IV over 30 minutes on Cycle 1 Day 1.
  Cycle 2 & Cycle 3 Day 1: Pembrolizumab 200 mg is administered by IV over 30 minutes
  Cycle 2 & Cycle 3 either Day 1 or Day 2 (within 36 hours of receiving pembrolizumab): patients undergo cryosurgery (injection of 30-60 x 10^6 mDCs and an injection of 0.5 ml Prenar13 such that two distinct metastatic lesions are cryoablated, one during cycle 2 and the other during cycle 3.
  Cycle 4 Day 1 and all subsequent cycles for a maximum of 2 years: Pembrolizumab 200 mg is administered by IV over 30 minutes
- Phase I Schedule 2: Cycle length is 21 days with the exception of cycle 1 which may be extended an additional 7 days to allow for dendritic cell production
  Patients undergo apheresis over 4 hours and pembrolizumab IV over 30 minutes on Cycle 1 Day 1.
  Cycle 2 & Cycle 3 Day 1 or Day 2: patients undergo cryosurgery (injection of 30-60 x 10^6 mDCs and an injection of 0.5 ml Prenar13 such that two distinct metastatic lesions are cryoablated, one during cycle 2 and the other during cycle 3.
  Cycle 4 Day 1 and all subsequent cycles for a maximum of 2 years: Pembrolizumab 200 mg is administered by IV over 30 minutes
Arm/Group | Phase I Schedule 1 | Phase I Schedule 2
Number analyzed (Participants) | 7 | 0
Participants
  Number of patients who developed a DLT on Schedule 1 | 0 | 0
  Number of patients who did not develop a DLT on Schedule 1 | 7 | 0

2. Secondary Outcome: Incidence of Adverse Events
Description: Assessed using Common Terminology Criteria for Adverse Events (CTCAE).
Time Frame: 30 months (through study completion)
Population: All patients who were eligible and started protocol treatment
Measure: Count of Participants; unit: Participants
Groups:
- Phase I Schedule 1: Cycle length is 21 days with the exception of cycle 1 which may be extended an additional 7 days to allow for dendritic cell production
  Patients undergo apheresis over 4 hours and pembrolizumab IV over 30 minutes on Cycle 1 Day 1 on day 1. ( Cycle 2 & Cycle 3 Day 1: Pembrolizumab 200 mg is administered by IV over 30 minutes
  Cycle 2 & Cycle 3 either Day 1 or Day 2 (within 36 hours of receiving pembrolizumab): patients undergo cryosurgery (injection of 30-60 x 10^6 mDCs and an injection of 0.5 ml Prenar13 such that two distinct metastatic lesions are cryoablated, one during cycle 2 and the other during cycle 3.
  Cycle 4 Day 1 and all subsequent cycles for a maximum of 2 years: Pembrolizumab 200 mg is administered by IV over 30 minutes
- Phase 1 Schedule -1: Cycle length is 21 days with the exception of cycle 1 which may be extended an additional 7 days to allow for dendritic cell production
  Patients undergo apheresis over 4 hours and pembrolizumab IV over 30 minutes on Cycle 1 Day 1.
  Cycle 2 & Cycle 3 Day 1: patients undergo cryosurgery (injection of 30-60 x 10^6 mDCs and an injection of 0.5 ml Prenar13 such that two distinct metastatic lesions are cryoablated, one during cycle 2 and the other during cycle 3.
  Cycle 4 Day 1 and all subsequent cycles for a maximum of 2 years: Pembrolizumab 200 mg is administered by IV over 30 minutes
Arm/Group | Phase I Schedule 1 | Phase 1 Schedule -1
Number analyzed (Participants) | 7 | 0
Participants
  grade 3 headache | 1 |
  grade 2 creatinine increase | 1 |
  grade 2 aspartate aminotransferase increase | 1 |
  grade 2 fatigue | 2 |
  grade 2 fever | 1 |
  grade 2 hyperglycemia | 2 |
  grade 2 pain | 2 |
  grade 3 hypertension | 1 |
  grade 2 blood bilirubin increase | 1 |

3. Secondary Outcome: Overall Survival
Description: Time from registration to death due to any cause
Time Frame: 30 months (through study completion)
Measure: Median (Full Range); unit: days
Groups:
- Treatment (Apheresis, Pembrolizumab, Cryosurgery, Mature Dendritic Cells [mDCs]): Cycle length is 21 days with the exception of cycle 1 which may be extended an additional 7 days to allow for dendritic cell production
  Patients undergo apheresis over 4 hours and pembrolizumab IV over 30 minutes on Cycle 1 Day 1 on day 1. ( If first mDC production attempt does not yield any releasable mDCs then one additional apheresis may be attempted.)
  Cycle 2 & Cycle 3 Day 1: Pembrolizumab 200 mg is administered by IV over 30 minutes
  Cycle 2 & Cycle 3 either Day 1 or Day 2 (within 36 hours of receiving pembrolizumab): patients undergo cryosurgery (injection of 30-60 x 10^6 mDCs and an injection of 0.5 ml Prenar13 such that two distinct metastatic lesions are cryoablated, one during cycle 2 and the other during cycle 3.
  Cycle 4 Day 1 and all subsequent cycles for a maximum of 2 years: Pembrolizumab 200 mg is administered by IV over 30 minutes
Arm/Group | Treatment (Apheresis, Pembrolizumab, Cryosurgery, Mature Dendritic Cells [mDCs])
Number analyzed (Participants) | 7
days | 211 [11 to 751]

4. Other Pre Specified Outcome: Progression-free Survival Time
Description: time from registration to disease progression (per RECIST criteria) or death due to any cause
Time Frame: 30 months (through study completion)
Population: The trial closed to enrollment following Phase I Schedule 1 testing due to poor accrual.
Measure: Median (Full Range); unit: days
Groups:
- Phase I Schedule 1: Cycle length is 21 days with the exception of cycle 1 which may be extended an additional 7 days to allow for dendritic cell production
  Patients undergo apheresis over 4 hours and pembrolizumab IV over 30 minutes on Cycle 1 Day 1 on day 1.
  Cycle 2 & Cycle 3 Day 1: Pembrolizumab 200 mg is administered by IV over 30 minutes
  Cycle 2 & Cycle 3 either Day 1 or Day 2 (within 36 hours of receiving pembrolizumab): patients undergo cryosurgery (injection of 30-60 x 10^6 mDCs and an injection of 0.5 ml Prenar13 such that two distinct metastatic lesions are cryoablated, one during cycle 2 and the other during cycle 3.
  Cycle 4 Day 1 and all subsequent cycles for a maximum of 2 years: Pembrolizumab 200 mg is administered by IV over 30 minutes
- Phase I Schedule -1: Cycle length is 21 days with the exception of cycle 1 which may be extended an additional 7 days to allow for dendritic cell production
  Patients undergo apheresis over 4 hours and pembrolizumab IV over 30 minutes on Cycle 1 Day 1.
  Cycle 2 & Cycle 3 Day 1: patients undergo cryosurgery (injection of 30-60 x 10^6 mDCs and an injection of 0.5 ml Prenar13 such that two distinct metastatic lesions are cryoablated, one during cycle 2 and the other during cycle 3.
  Cycle 4 Day 1 and all subsequent cycles for a maximum of 2 years: Pembrolizumab 200 mg is administered by IV over 30 minutes
- Phase II Schedule: Phase II Schedule depends on the Phase I findings
Arm/Group | Phase I Schedule 1 | Phase I Schedule -1 | Phase II Schedule
Number analyzed (Participants) | 7 | 0 | 0
days | 88 [11 to 113] |  |

ADVERSE EVENTS:
Time Frame: 30 months (through study completion)
Description: CTCAE criteria grade 2 or higher regardless of attribution
Groups:
- Phase I Schedule -1: Phase I Schedule -1 Treatment cohort where cycle length is 21 days: On D1C1, patients undergo apheresis and receive 200mg pembrolizumab IV over 30 minutes. On C2D1, a single metastatic lesion will be biopsied and cryoablated (using conventional freeze-thaw-freeze cycle). After the lesion has thawed, a 22 G needle will be placed under ultrasound or CT-guidance into the ablated portion of the lesion. The mature Dendritic Cells (total mDCS: 30-60 x10^6) will be administered through this needle over different areas of the cryoablated region and then flushed with 1ml of sterile saline. Prevnar13® will be injected into the ablated portion of the lesion after administration of mDCs. On C3D1 the same treatment will be administered to a different metastatic lesion. C4D1 and D1 of all subsequent cycle patients will receive 200mg pembrolizumab IV over 30 minutes. Treatment continues until disease progression or a maximum of 24 months post registration.
- Phase II Schedule: Phase II schedule depends on the result of the Phase I portion of the study
Arm/Group | Phase I Schedule 1 | Phase I Schedule -1 | Phase II Schedule
All-Cause Mortality (participants affected / at risk) | 7/7 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 2/7 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 4/7 | 0/0 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase I Schedule 1 (N=7) | Phase I Schedule -1 (N=0) | Phase II Schedule (N=0)
grade 3 hypertension (Vascular disorders) | 1 | 0 | 0
grade 3 headache (Nervous system disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Phase I Schedule 1 (N=7) | Phase I Schedule -1 (N=0) | Phase II Schedule (N=0)
Grade 2 blood bilirubin increase (Investigations) | 1 | 0 | 0
Grade 2 Aspartate aminotransferase increased (Investigations) | 1 | 0 | 0
Grade 2 Creatinine increase (Investigations) | 1 | 0 | 0
Grade 2 fatigue (General disorders) | 2 | 0 | 0
Grade 2 fever (General disorders) | 1 | 0 | 0
Grade 2 pain (General disorders) | 2 | 0 | 0
Grade 2 hyperglycemia (Metabolism and nutrition disorders) | 2 | 0 | 0

LIMITATIONS AND CAVEATS:
The trial was closed to enrollment during the Phase I portion of the trial due to poor enrollment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-07-03): https://cdn.clinicaltrials.gov/large-docs/01/NCT03325101/Prot_SAP_000.pdf
  • Informed Consent Form (2020-07-17): https://cdn.clinicaltrials.gov/large-docs/01/NCT03325101/ICF_001.pdf